CLINICAL TRIAL: NCT03036358
Title: The Effect of Teledermatology on Length of Hospital Admission, Length of Stay, 30 Day Readmission Rate, and Antibiotic Use in Patients Presenting With Cellulitis vs Pseudocellulitis in an Academic Emergency Department Setting.
Brief Title: Effect of Teledermatology on Length of Hospital Admission, Length of Stay, 30 Day Readmission Rate, and Antibiotic Use in Patients Presenting With Cellulitis vs Pseudocellulitis in an Academic ED Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Benjamin Kaffenberger, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2015H0134
Record Dates: First submitted 2016-06-04; First posted 2017-01-30 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Cellulitis
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teledermatology consult (Other): To determine the benefit of teledermatology to differentiate cellulitis from pseudocellulitis in emergency departments through the analysis of time spent in the emergency department (ED), admission to the inpatient hospital, antibiotic use, time to improvement, and 30-day remission rate. This arm will undergo imaging, a dermatologic assessment will be performed, AND this assessment will be entered into the patients chart.
  Interventions: Other: teledermatology consult
- Routine Care (Other): To determine the benefit of teledermatology to differentiate cellulitis from pseudocellulitis in emergency departments through the analysis of time spent in the emergency department (ED), admission to the inpatient hospital, antibiotic use, time to improvement, and 30-day remission rate. This arm will undergo imaging, a dermatologic assessment will be performed, AND this assessment WILL NOT be entered into the patients chart
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: teledermatology consult — Information from the dermatologic assessment will be entered into the patients chart.
  Arms: Teledermatology consult
Other: Routine Care — The dermatologic assessment will occur but not added to the patients medical record. Dermatology may still be consulted but will be at the prerogative of the treating hospitalist.
  Arms: Routine Care

SUMMARY:
The effect of teledermatology on length of hospital admission, length of stay, 30 day readmission rate, and antibiotic use in patients presenting with cellulitis vs pseudocellulitis in an academic emergency department setting.

DETAILED DESCRIPTION:
The Investigator hope to determine if the implementation of teledermatology in the emergency department (ED) at The Ohio State University Wexner Medical Center is beneficial in diagnosing cases of cellulitis and pseudocellulitis conditions. Prior studies have indicated that misdiagnosis may occur in up to 28% of patients in the ED with these conditions. Additionally, dermatological consults have been shown to change diagnosis or management of these conditions in more than 60% of the patients examined. Without the use of teledermatology, however, a dermatological consult would be prohibitively expensive and take time to obtain. The investigator proposes that by utilizing teledermatology in emergency rooms, the investigator can make faster, yet just as accurate, dermatological diagnoses in patients presenting with cellulitis-like symptoms. Subsequently, by reducing the number of misdiagnoses, unnecessary use of antibiotics and hospitalizations will also decrease, lowering health care costs and simultaneously providing patients with faster treatment of the actual dermatologic condition.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Present to the ED with cellulitis-like symptoms, including but not limited to the following: tenderness, redness, swelling, expansive lesion

Exclusion Criteria:

* pregnant
* prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Admission to the hospital | 30 days
  To determine the benefit of teledermatology to differentiate cellulitis from pseudocellulitis in emergency departments through the analysis of time spent in the emergency department (ED), admission to the inpatient hospital, antibiotic use, time to improvement, We anticipate a high rate of pseudocellulitis, and this aim will determine if there is a difference in patient admissions among those who receive a dermatologic assessment

SECONDARY OUTCOMES:
Length of stay in the hospital | 30 days post admission
  Will assess time spent in the hospital for those that were admitted
30 day readmission rate | 30 days post admission
  Will assess hospitalization/emergency department readmission in the following 30 days
Antibiotic use | 30 days post admission
  Will assess the frequency of antibiotic use between groups

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Kaffenberger, MD, Principal Investigator — OSU Dermatology
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes